CLINICAL TRIAL: NCT04418076
Title: Improving Antiretroviral Adherence and Persistence Using mHealth Tools in HIV-infected Cocaine Users
Brief Title: Project SMART Automated Pillbox Study
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University at Albany (Other); University of Connecticut (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1508016342; 1R21DA039842-01A1 (NIH)
Record Dates: First submitted 2018-03-16; First posted 2020-06-05 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS; Cocaine Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- No feedback (Experimental): For participants in the control group (Group A), no feedback from the TowerView Health® smart pill box or clinical nurse will be given.
  Interventions: Device: Group A_No feedback
- Automated feedback (Experimental): For participants in Group B (automated feedback), automated feedback will be generated from the TowerView Health® smart pill box and sent to participants' smartphone as text messages.
  Interventions: Device: Group B_Automated feedback
- Automated feedback + Clinician feedback (Experimental): For participants in Group C, automated feedback will be generated from the TowerView Health® smart pill box and sent to participants' smartphone as text messages. In addition, clinical nurse will also send personalized feedback and suggestions to the participants in this group.
  Interventions: Device: Group C_Automated feedback + Clinician feedback
- Automated feedback + Social Network feedback (Experimental): For participants in Group D, automated feedback will be generated from the TowerView Health® smart pill box and sent to participants' smartphone as text messages. In addition, a weekly text reminder will be sent to each participant from a social network designee chosen by the participant.
  Interventions: Device: Group D_Automated feedback + Social Network feedback

INTERVENTIONS:
Device: Group A_No feedback — In the control (Group A), the feedback option will be deactivated on the device on the TowerView Health® smart pill box, effectively serving to only monitor natural pill-taking patterns.
  Arms: No feedback
Device: Group B_Automated feedback — For participants in Group B (automated feedback), missed dosages will prompt an automated text message to be sent to the participants' smartphone. The TowerView Health® pill box consists of in-built alarm and flashing color lights, and the ability to send text messages to the participants' phone either as reminder in the event of missed dosage or a message of encouragement when all dosages are taken.
  Arms: Automated feedback
Device: Group C_Automated feedback + Clinician feedback — For participants in Group C, the survey app responses will be assessed each week by the RA who in turn will communicate the results to a clinical nurse. The clinical nurse will be funded through this study; he/she will be responsible for providing personalized feedback to all Group C participants. The clinic nurse will contact the subject with appropriate feedback about their health behavior and suggestions for sustained adherence.
  Arms: Automated feedback + Clinician feedback
Device: Group D_Automated feedback + Social Network feedback — For participants in Group D, a social network designee will be chosen based on the names provided by the participants during screening. One social network designee will be consented and chosen to send the participant a weekly text reminder the participant to take their medication. The text for the message will be chosen by the social network designee.
  Arms: Automated feedback + Social Network feedback

SUMMARY:
The aim of this study is to examine the effect of mHealth tools on antiretroviral (ART) adherence and persistence among HIV-infected individuals with co-occurring cocaine use disorders (CUDs).

DETAILED DESCRIPTION:
To conduct qualitative assessments using focus groups of people living with HIV (PLH) who use cocaine and healthcare providers that will assess the acceptability, feasibility, facilitators and barriers of implementing mHealth interventions; and will aid in developing the final design and content of both automated and clinician feedback in preparation for designing a pilot feasibility study.

To conduct a 12-week pilot feasibility RCT among PLH with co-occurring CUDs that will examine the impact of mHealth tools (cellular-enabled smart pill boxes and cell phones) and feedback (no feedback vs. automated feedback vs. automated + clinician feedback) on primary (ART adherence and persistence) and secondary outcomes (HIV viral suppression, cocaine use, retention in HIV care).

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Clinic-confirmed HIV diagnosis
* Currently prescribed or eligible for ART
* Currently has insurance
* Self-reported cocaine use in the past 30 days
* Willing and able to use a cell phone and electronic pill box for the 12-week intervention

Exclusion Criteria:

* Unable to provide informed consent
* Verbally or physically threatening to research staff
* Unable to communicate in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, M.D., M.A., Principal Investigator — Yale University
Locations (1):
- Yale Clinical Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
All data will be kept confidential.

REFERENCES:
- [Derived] Ranjit YS, Krishnan A, Ghosh D, Cravero C, Zhou X, Altice FL. mHealth Intervention to Improve Treatment Outcomes Among People With HIV Who Use Cocaine: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 7;11(3):e28332. doi: 10.2196/28332. PMID 35254270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two sites--New Haven and Hartford, CT. Recruitment started in June 2017 and concluded in January 1st 2020.
Pre-assignment Details: This study required participants to change their pharmacy for delivery of HIV medication , so that the medication blister pack could be inserted into the TowerView smart pillbox. In some cases, participants who had severe opioid use disorder were prevented by their provider from participating in this study; they prefer close monitoring. Other factors preventing participants from continuing included co-morbidities (cancer, severe SUD), incarceration, and difficulty with transportation.
Period: Overall Study
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Started | 19 | 20 | 16 | 23
9 Participants Had Complete Lab Results at 16 Weeks | 1 | 3 | 4 | 1
57 Participants Completed 12 Weeks | 15 | 15 | 11 | 16
Completed | 13 | 15 | 12 | 17
Not Completed | 6 | 5 | 4 | 6
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 5 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Dropped out after receiving pillbox and phone | 2 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback | Total
Number analyzed (Participants) | 19 | 20 | 16 | 23 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.91 (7.70) | 54.78 (6.81) | 51.45 (6.45) | 55.94 (6.35) | 54.65 (6.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 8 | 6 | 13 | 39
  Female | 7 | 9 | 9 | 9 | 34
  Transgender (male to female) | 0 | 3 | 1 | 1 | 5
  Transgender (female to male) | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 5 | 2 | 18
  Black | 10 | 13 | 10 | 17 | 50
  Hispanic or Puerto Rican | 3 | 2 | 1 | 4 | 10
Health literacy [Mean (Standard Deviation); unit: units on a scale] — It includes three Likert scale questions on a scale of 1 to 5. The scores of each question were averaged to obtain an average score. Higher score indicates higher level of health literacy.
  units on a scale | 4.04 (.99) | 3.92 (.92) | 3.92 (.85) | 3.86 (1.02) | 3.93 (.94)
Mental health (CESD-D10) [Mean (Standard Deviation); unit: units on a scale] — The CES-D Scale: A self-report depression scale for research in the general population. It includes 10 questions, measured from 0 to 3, where higher score indicates higher level of depression. All of the questions are totaled, thus minimal is 0 and maximum is 30.
  units on a scale | 10.89 (6.67) | 9.80 (7.13) | 9.56 (6.18) | 11.43 (7.20) | 10.50 (6.77)
Alcohol screening AUDIT C [Mean (Standard Deviation); unit: units on a scale] — Scales measure substance use using multiple choices. Questions were coded as 0, 1 to 4. The results were summed up for each participant. If the sum >=2, then presence of substance use, else no substance use. Answers are summed up, 0 is the minimal and 12 is the maximum.
  units on a scale | 5.50 (3.09) | 3.46 (3.13) | 5.10 (3.64) | 4.00 (2.88) | 4.45 (3.17)
Presence of cocaine use disorder [Count of Participants; unit: Participants]
  Yes | 19 | 19 | 16 | 21 | 75
  No | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Anti-Retroviral Therapy (ART) at the End of 12-Week Intervention Period
Description: Adherence will be measured in percentage of times pills taken in time or within 90 mins of reminder based on the real time record of the behavior provided by the electronic pill box.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: percentage of times pills taken
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Number analyzed (Participants) | 15 | 15 | 11 | 16
percentage of times pills taken | 91.07 (25.58) | 96.00 (12.98) | 99.82 (.60) | 94.81 (13.48)

2. Primary Outcome: Adherence to Anti-Retroviral Therapy (ART) at the End of 16 Weeks (4-week Post-intervention Period)
Description: This is a follow up period where participants adherence will be measured in percentage of times pills taken in time or within 90 mins of reminder after being the study for 16 weeks. The information will be based on the real time record of the behavior provided by the electronic pill box.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: percentage of times pills taken
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Number analyzed (Participants) | 13 | 15 | 12 | 17
percentage of times pills taken | 96.31 (7.49) | 93.00 (25.76) | 92.75 (21.53) | 93.24 (24.15)

3. Secondary Outcome: Changes in HIV 1 RNA, QN PCR (Copies/ML)
Description: HIV RNA (viral load) and HIV disease progression to manage and monitor HIV infection.
Time Frame: End of intervention (Week 12)
Population: If there is a change from viral suppression or not viral suppression to maximum viral suppression between baseline and intervention end date. Maximum viral suppression is <20, viral suppression is <200, not viral suppression is >200 copies/ML. Only 26 participants whose labs are complete. Thus we were only able to analyze this outcome on 26 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Number analyzed (Participants) | 8 | 10 | 8 | 0
Participants
  Changed to maximum viral suppression | 0 | 2 | 2 |
  Viral load decreased but not achieve max viral suppression | 0 | 0 | 2 |
  Viral load increase | 3 | 3 | 1 |
  No change and remained max suppression | 5 | 4 | 3 |
  No change and remained viral suppression or no viral suppression | 0 | 1 | 0 |

4. Secondary Outcome: Percent Change in CD4 Count From Baseline to Week 12
Description: CD4 T lymphocyte (CD4) cell count are markers of antiretroviral treatment (ART) responses. Participants will be asked to perform testing including CD4 lymphocyte count at the end of intervention (Week 12). The value is calculated by the percentage of CD4 at Week 12 minus the percentage of CD4 at baseline.
Time Frame: Baseline and End of intervention (Week 12)
Population: 18 lab results were missing or lost and not available. 60 participants submitted their CD4 data (summarized here) vs. 57 participants completed all data measures at week 12.
Measure: Mean (Standard Deviation); unit: percentage of CD4 (helper cells)
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Number analyzed (Participants) | 14 | 15 | 14 | 17
percentage of CD4 (helper cells) | 27.00 (13.33) | 26.09 (12.75) | 28.8 (9.96) | 30.81 (6.56)

5. Secondary Outcome: Retention in Care
Description: Participants medical chart review will be reviewed to look at the number of doctor's visit for for the duration of the study (4 months).
Time Frame: up to End of the study (week 16)
Population: These data were not collected due to changes in the research plan.
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | No Feedback | Automated Feedback | Automated Feedback + Clinician Feedback | Automated Feedback + Social Network Feedback
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/20 | 0/16 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/16 | 0/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/16 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT04418076/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04418076/ICF_001.pdf